CLINICAL TRIAL: NCT05948345
Title: Exploring the Real-life Stories of Individuals Enrolled in Lymphedema Clinical Trials
Brief Title: Evaluating Factors In Study Experiences of Lymphedema Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83474689
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lymphedema
Keywords: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study intends to investigate the personal experiences of lymphedema patients who take part in a separate clinical trial including a specific medication intervention. The major focus will be on closely following individuals' rates of trial completion and withdrawal.

The data collected from this study will help improve future outcomes for all lymphedema patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lymphedema
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphedema who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a lymphedema clinical trial | 3 months
Rate of patients who remain in lymphedema clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quere I, Presles E, Coupe M, Vignes S, Vaillant L, Eveno D, Laporte S, Leizorovicz A; POLIT Study investigators. Prospective multicentre observational study of lymphedema therapy: POLIT study. J Mal Vasc. 2014 Jul;39(4):256-63. doi: 10.1016/j.jmv.2014.05.004. Epub 2014 Jun 12. PMID 24931830
- [Background] Boccardo F, Santori G, Villa G, Accogli S, Dessalvi S. Long-term patency of multiple lymphatic-venous anastomoses in cancer-related lymphedema: A single center observational study. Microsurgery. 2022 Oct;42(7):668-676. doi: 10.1002/micr.30944. Epub 2022 Aug 2. PMID 35916247
- [Background] Johansson K, Blom K, Nilsson-Wikmar L, Brogardh C. Early Intervention with a Compression Sleeve in Mild Breast Cancer-Related Arm Lymphedema: A 12-Month Prospective Observational Study. Cancers (Basel). 2023 May 9;15(10):2674. doi: 10.3390/cancers15102674. PMID 37345010

DOCUMENTS (1):
  • Informed Consent Form (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT05948345/ICF_000.pdf